CLINICAL TRIAL: NCT00011089
Title: US Expanded Access Program of Tenofovir Disoproxil Fumarate in the Treatment of HIV-1 Infected Patients Who Have Limited Treatment Options
Brief Title: Tenofovir Disoproxil Fumarate in HIV-Infected Patients Who Have Not Had Success With Other Anti-HIV Drug Combinations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 283G; GS-00-955
Record Dates: First submitted 2001-02-09; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-11

CONDITIONS: HIV Infections
Keywords: HIV-1; Disease Progression; Reverse Transcriptase Inhibitors; Anti-HIV Agents; 9-(2-phosphonylmethoxypropyl)adenine
MeSH Terms: conditions — HIV Infections; Disease Progression | interventions — Tenofovir

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate

SUMMARY:
The purpose of this study is to make tenofovir disoproxil fumarate (DF) available to HIV-infected patients who have failed other anti-HIV drug combinations, who have few treatment choices available, and whose disease may get worse. This study will allow patients to obtain tenofovir DF before it is approved for marketing.

DETAILED DESCRIPTION:
Patients receive daily doses of tenofovir DF.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have a viral load (level of HIV in the blood) of at least 10,000 copies/ml by PCR within the previous 2 months.
* Have a CD4 count of 100 cells/mm3 or lower within the previous 2 months. Patients with a CD4 count above 100 and as high as 200 cells/mm3 may also be eligible if they had an opportunistic (AIDS-related) infection within the past 90 days.
* Have failed treatment with at least 2 protease inhibitors (PIs) or at least 1 PI plus a nonnucleoside reverse transcriptase inhibitor (NNRTI).
* Are not able to get effective treatment with a combination of currently approved anti-HIV drugs.
* Are at least 18 years old.
* Have a negative serum pregnancy test.
* Are willing to use a barrier method of birth control (both males and females) while on the study and for 30 days after taking the drug.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have or have had kidney disease or bone disease.
* Are pregnant or breast-feeding.
* Abuse alcohol or drugs.
* Are taking, or have taken within 7 days of enrolling in the study, adefovir dipivoxil or drugs that may cause kidney problems, including aminoglycoside antibiotics, cidofovir, foscarnet, intravenous (IV) amphotericin B, IV pentamidine, IV vancomycin, and chemotherapy (e.g., cisplatin).
* Have any medical conditions or have had any medications that the study investigator believes will make him/her unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-02

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Information, Foster City, California, United States